CLINICAL TRIAL: NCT03832140
Title: Frequency and Characteristics of Pruritus in Patients With Monoclonal Gammopathy
Acronym: PRURIGAMMA
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PRURIGAMMA (29BRC18.0192)
Record Dates: First submitted 2019-02-05; First posted 2019-02-06 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Pruritus; Monoclonal Gammopathy
MeSH Terms: conditions — Pruritus; Paraproteinemias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with monoclonal gammopathy
- patients with a normal plasma protein electrophoresis

SUMMARY:
Pruritus is most often secondary to dermatitis but can also occur without skin lesions, it is called pruritus sine materia. The causes of pruritus sine materia are various: haematological (myeloproliferative neoplasia ...), hepatic (cholestasis ...), renal (chronic renal failure, dialysis), endocrine (iron deficiency ...), secondary to drug intake ... or idiopathic when no cause is found.

Gammapathies are among the causes of pruritus sine materia, and as such electrophoresis of serum proteins is usually part of the pruritus assessment to look for monoclonal gammopathy (MGUS, multiple myeloma, Waldenström disease). However, there is very little data on the frequency of pruritus in patients with monoclonal gammopathy and the characteristics of this pruritus. So the aim of this study is to compare the frequency of pruritus between patients with monoclonal gammapathy and controls

ELIGIBILITY:
Inclusion Criteria for case :

Major patient Realized Serum protein electrophoresis between 2014 and 2017 Hematology follow-up at Brest CHR Positive monoclonal gammopathy Non-opposition formulated

Inclusion Criteria for Control :

Major patient Realized Serum protein electrophoresis between 2014 and 2017 Hematology follow-up at Brest CHR Negative gammopathy Non-opposition formulated

Exclusion Criteria:

Minor patient Major protected Patient with another haemopathy secreting a monoclonal immunoglobulin (lymphoma, LLC ...) Physical or mental incapacity Refusal to participe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had serum protein electrophoresis at Brest CHRU between 2014 and 2017, with and without gammapathy.
Sampling Method: Non-Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-11-19 (Actual)

PRIMARY OUTCOMES:
Frequency of pruritus | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending three years maximum following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. requestors will be required to sign and complete a data access agreement